CLINICAL TRIAL: NCT04234737
Title: Efficacy of Hypnotherapy in Children Aged 8-12 Years Old With Dental Anxiety: A Randomized Clinical Trial
Brief Title: Efficacy of Hypnotherapy in Children With Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Kardes, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 352684
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; hypnotherapy; pediatric dentistry
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotherapy (Experimental)
  Interventions: Behavioral: Hypnotherapy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Hypnotherapy — Hypnotherapy
  Arms: Hypnotherapy

SUMMARY:
Dental anxiety is a common problem among the children. The aim of this study is to evaluate the efficacy of hypnotherapy in children with dental anxiety. The participants will be randomized in a 1:1 ratio to hypnotherapy or control group. The outcome measures will be Modified Children Dental Anxiety Scale-faces version(MCDAS(f)) and Visual Analogue Scale(VAS).

ELIGIBILITY:
Inclusion Criteria:

* initial MCDAS(f) total score > 19
* ICDAS II (international caries detection and assessment score)= 5 for at least one tooth

Exclusion Criteria:

* presence of dental pain complaint
* non-obtaining the informed consent form

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Modified Children Dental Anxiety Scale Faces version MCDAS(f) | maximum 1 week after hypnotherapy.
  Modified Children Dental Anxiety Scale is a self-reported measurement and consists of 8 questions with 5 pictorial answers for each question. Total score ranges from 8 to 40, with higher scores higher dental anxiety.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | during dental treatment
  Visual Analog Scale was used to evaluate the dental anxiety in six stages of dental treatment. The scores range from 0 to 10, with higher scores higher dental anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Sengul, Study Director — assistant professor
Locations (1):
- Ataturk University Faculty of Dentistry Pediatric Dentistry Department, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided